CLINICAL TRIAL: NCT00564200
Title: MINIALO-VELCADE2005: A Phase II National, Open-label, Multicenter, no Controlled Study of Treated With Bortezomib (Velcade) Multiple Myeloma Patients Pre and Post Allogeneic Haematopoietic Progenitor Cell Transplant With no Myeloablative Conditioning
Brief Title: MINIALO-VELCADE2005: A Study of Bortezomib (Velcade) Treated Multiple Myeloma Patients Pre and Post Allogeneic Haematopoietic Progenitor Cell Transplant With no Myeloablative Conditioning
Acronym: MINIALO-VELCAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-004858-27
Record Dates: First submitted 2007-11-26; First posted 2007-11-27 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma, transplant
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Dexamethasone; fludarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Bortezomib — PREACONDICIONAMIENTO:
  * 2 cycles of 21 days : Velcade days: 1, 4, 8 and 11
  * 1 cycle of 13 days : Velcade days 1, 4, 8 and 11
  ACONDICIONAMIENTO:
  - Day -2: Velcade
  POSTRANSPLANTATION:
  * 2 cycles of 21 days : Velcade days 1, 8 and 15
  * 5 cycles of 56 days : Velcade days 1, 8 and 15
Drug: dexamethasone — PREACONDICIONAMIENTO:
  - 2 cycles of 21 days : Dexamethasone: days 1-4 and 8-11
Drug: Fludarabine — ACONDICIONAMIENTO:
  - Days -9 al -5: Fludarabine
Drug: Melphalan — ACONDICIONAMIENTO:
  - Days -4 and -3: Melphalan.

SUMMARY:
The primary objective of this study is to analyze the efficacy of allogeneic bone marrow transplantation in a reduced-intensity manner combined with bortezomib in the treatment of multiple myeloma with bad prognosis, in order to evaluate the response and relapse rates

DETAILED DESCRIPTION:
Multiple Myeloma is a plasma cell disorder characterized by an uncontrolled proliferation of bone marrow plasma cells leading to skeletal destruction with bone pain, anemia, renal failure, hypercalcemia, recurrent bacterial infections and extramedullary plasmacytomas. It accounts for 1% of all malignancies and slightly more than 10% of hematologic malignancies, with an annual incidence of about four per 100.000. Although this disease is incurable with a median survival of about 3 years, remarkable treatment advances have been recently made, including high-dose therapy followed by stem cell rescue and, particularly, the introduction of novel promising agents with new mechanisms of action.

The treatment with alquilant agents, melphalan or cyclophosphamide combined with prednisone has a median of no more than 3 years survival rate in approximately 50%. The chemotherapy combination and high-dose dexamethasone increases response rate with minimal effects in survival benefit. The limited efficacy of conventional treatment produced the introduction of the high-dose therapy followed by a stem cells transplant in order to increase antitumoral effect and prolong disease-free overall survival.

This way, autologous stem cells transplant has turned into optimal treatment for patients younger than 65 years with myeloma. Nevertheless there is increasing evidence that it benefits only patients who showed complete disease remission after transplantation.

The transcendental factor that determines the CR post-transplantation achievement is the initial chemotherapy- sensitivity disease, measuring the rapidity and the grade of response (rapidity of maximum response assessment) and the pre-transplantation M protein level (i.e., the grade of response to the initial treatment).

On the other hand, the treatments with alquilant agents can impede the obtention of adequate numbers of stem cells that make impossible the autotransplantation practice. For this reason nowadays the treatments based on dexamethasone are used as initial chemotherapy.

However, these regimens and particularly AVD have less activity than alquilant agents treatment. Bortezomib has shown a fast antimyeloma activity (response after 1 or 2 cycles) in refractory patients, where myelosuppression and cellular injury are not observed.

Alternating bortezomib and dexamethasone as pre-transplant induction regimen would show the following advantages:

1. a rapid and high effect raised by means of the use of two drugs with proven activity when they are administered separately,
2. absence of stem cells injury,
3. different toxicity types avoiding the habitual side effects because of the dexamethasone abuse, when this one is administered in every cycle as it happens in AVD type regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patient is, in the investigator's opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Age over 18 and under 67 years old.
* Patient diagnosed with symptomatic Multiple Myeloma based on standard criteria with bad prognosis. This factor is associated with at least one of the clinical alterations defined as follows:

Patient who displayed a Monosomy of chromosome 13 or other adverse cytogenetic abnormality.

Patient in first relapse. Patient with relapsed multiple myeloma after autologous transplantation.

* Patient has a ECOG performance status <= 2.
* Patient has a life-expectancy >3 months.
* Patients who are candidates for autologous transplantation.
* Patients must have HLA-identical sibling donors.
* Patient has the following laboratory values before Baseline visit:

Platelet count ≥ 30000/mm3 (transfusion allowed), hemoglobin ≥ 8 g/dl (transfusion allowed) and absolute neutrophil count (ANC) ≥ 0.750/mm3. Lower values are accepted if they are caused by bone marrow infiltration.

Aspartate transaminase (AST): ≤ 2.5 x the upper limit of normal. Alanine transaminase (ALT): ): ≤ 2.5 x the upper limit of normal. Total bilirubin: ≤1.5 x the upper limit of normal. Serum creatinine value ≤ 2mg/dl

Exclusion Criteria:

* Patient present serious pathologies that make impossible chemotherapy treatments:

  1. Congestive heart failure, angina or heart attack during last 12 months.
  2. Uncontrolled arterial hypertension.
  3. Uncontrolled supraventricular arrhythmias during last 3 last months.
  4. Ventricular arrhythmia.
  5. Hepatic disease (Cirrhosis).
* Patient has Grade 2 peripheral neuropathy within 14 days before enrollment.
* Patient with serious psychiatric disorders that make impossible comply satisfactorily with the protocol requirements.
* Personal medical history of neoplasia of other type, except: carcinoma in situ, other curatively treated malignancy in complete remission for more than 10 years.
* Patient has hypersensitivity to bortezomib, boron or mannitol.
* Fertile patient is not going to use a medical effective contraceptive method during the trial.
* Patient has received other investigational drugs within 30 days before enrollment
* Patient is known to be seropositive for the human immunodeficiency virus (HIV), Hepatitis B surface antigen-positive or active hepatitis C infection.
* Patient had a myocardial infarction within 6 months of enrollment or has New York Heart Association (NYHA) Class III or IV, heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Patient is enrolled in another clinical research study and/or is receiving an investigational agent for any reason.
* Patient participated in clinical study VISTA.
* Pregnant or breast-feeding women.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-11; Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Analyze the efficacy of allogeneic bone marrow transplantation in a reduced-intensity manner combined with bortezomib | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bladé Joan, Dr, Study Chair — Hospital Clinic of Barcelona
Locations (10):
- Spain (10):
  - H. Clinic I Provincial, Barcelona
  - H. de la Santa Creu I Sant Pau, Barcelona
  - Instituto Catalán de Oncología, Barcelona
  - H. de Jerez, Jerez de la Frontera
  - H. 12 de Octubre, Madrid
  - H. Univ. Gregorio Marañón, Madrid
  - H. Univ. La Princesa, Madrid
  - H. Univ. Morales Meseguer, Murcia
  - H. Univ. Son Dureta, Palma de Mallorca
  - H. Univ. de Salamanca, Salamanca

REFERENCES:
- See also: Spanish association of Haematology — http://www.aehh.org